CLINICAL TRIAL: NCT05753384
Title: Discontinuation of TyrosIne Kinase Inhibitors (ITK) in Chronic Myeloid Leukemia (LMC) and Impact on the Immune System: a Randomized Comparative Study of Two Therapeutic Strategies
Brief Title: Discontinuation of TyrosIne Kinase Inhibitors (TKI) in Chronic Myeloid Leukemia (CML) and Impact on the Immune System
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AITIK
Record Dates: First submitted 2023-02-09; First posted 2023-03-03 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Tyrosine Kinase Inhibitors; Chronic Myeloid Leukemia
Keywords: Characteristics of innate T cells
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- continued treatment with TKI at 50% dose reduction (Experimental): continued treatment with TKI at 50% dose reduction compared to dosing received at randomization and then stopped treatment 12 months after randomization
  Interventions: Drug: treatment of TKI in CML
- continuation of TKI treatment without dose change (Active Comparator): continued treatment with TKI at same dose compared to dosing received at randomization and then stopped treatment 12 months after randomization
  Interventions: Drug: treatment of TKI in CML

INTERVENTIONS:
Drug: treatment of TKI in CML — continued treatment with TKI at randomization a then stopped treatment 12 months after randomization

SUMMARY:
Tyrosine kinase inhibitors (TKI) have revolutionized the management and prognosis of chronic myeloid leukemia (CML). Daily treatment with TKI, which is necessary due to lack of cure, is frequently associated with moderate, chronic and sometimes severe adverse effects. The ability to permanently stop treatment with TKI has thus become a major goal in CML to prevent the occurrence of adverse events, improve quality of life and reduce the general cost of the treatment; we talk about Treatment Free Remission (TFR). It now remains to be demonstrated in a comparative prospective study that a strategy of de-escalation of the TKI treatment dose before treatment discontinuation optimizes TFR results. At the same time, it is possible to reduce adverse reactions and improve the quality of life of patients. In this context, the investigator propose to conduct a randomized clinical trial including CML patients, allowing to compare the results of TFR at 24 months between a sudden stop of treatment after a maintenance phase of dosage for 12 months and a de-escalation arm of dose (dosage reduced by 50%) for 12 months before stopping. A secondary immunological translational objective of this project will be to compare the quantitative and qualitative evolution of innate CD8 T cells between the 2 arms (abrupt cessation of ITK treatment versus progressive withdrawal) and look for a predictive innate CD8 T cells blood signature at the time of stopping treatment of a successful TFR in both arms.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 year-old.
* Diagnosis of chronic phase CML according to WHO 2016 criteria with a typical BCR::ABL1 rearrangement (e13a2 or e14a2)
* Duration of treatment by Imatinib ≥ 4 years / ITK2G ≥ 3 years /Imatinib and ITK2G ≥ 4 years and no change of TKI or decrease in dosage in the last 6 months prior to inclusion
* Deep Molecular Response (DMR) duration ≥ 1 year
* Absence of contraindication to the continuation of the same TKI for 12 months at the same dosage according to international recommendations nd the PCR of each TKI:

Imatinib (≥ 300 mg/j) Dasatinib (≥ 50 mg/j) Nilotinib (≥ 300 mg/j) Bosutinib (≥ 200 mg/j)

* Patient not participating in another interventional study for the duration of the interventional study
* Sexually active men should use effective contraception when taking Dasatinib
* Having an health insurance
* Having signed the consent form

Non-Inclusion Criteria:

* Patients with progressive severe pathology of poor prognosis immediately compromising participation in the entire study and/or with uncontrolled chronic pathology
* ECOG ≥ 3
* Prior resistance to TKI
* Patients who have already experienced an attempt of TKI cessation
* Patients with a malignant tumour that has been treated with chemotherapy within 2 months of inclusion or undergoing chemotherapy or that will be treated with post-inclusion chemotherapy
* Protected person
* Pregnant women or women of childbearing age without appropriate contraceptive measures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2028-12-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients in treatment free Remission (TFR) 24 months after treatment discontinuation in patients.Treatment-Free Remission (TFR) is defined as patients with Major Molecular Response (MMR) or better (BCR-ABL level ≤ 0.1% IS). | 24 months after treatment discontinuation
  Percentage of patients in treatment free Remission (TFR) 24 months after treatment discontinuation in patients is calculated by dividing the number of patients with no loss of MMR-Major Molecular Response (BCR-ABL level ≤ 0.1% IS) on the total number of patients.

SECONDARY OUTCOMES:
Difference in proportions (%) at randomization and 12 months post randomization, of innate CD8 T cells among total CD8 T cells | 12 months

CONTACTS AND LOCATIONS:
Locations (20):
- France (20):
  - Chu Angers, Angers
  - Ch Annecy, Annecy
  - Ch Bayonne, Bayonne
  - Chu Brest, Brest
  - CH Brive la Gaillarde, Brive-la-Gaillarde
  - Ch Chambery, Chambéry
  - CHI Creteil, Créteil
  - Ch La Rochelle, La Rochelle
  - Chu Lille, Lille
  - CHU Limoges, Limoges
  - Centre Léon Bérard, Lyon
  - Ch Mont de Marsan, Mont-de-Marsan
  - Chu Nancy, Nancy
  - Chu Nantes, Nantes
  - Hopital Prive Du Confluent, Nantes
  - Ch Perigueux, Périgueux
  - Chu Poitiers, Poitiers
  - Oncopole Toulouse, Toulouse
  - Chu Tours, Tours
  - CH Versailles, Versailles